CLINICAL TRIAL: NCT01837017
Title: Project FARMS: Fall Risk Reduction in Multiple Sclerosis
Acronym: FARMS-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CMSC-2012; CMSC 2011-06476 (Other Grant/Funding Number: Consortium of Multiple Sclerosis Centers)
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Sclerosis
Keywords: Falls,; Balance,; Gait,; Older adults
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home-based Exercise (Experimental): The home-based exercise group attends 4 exercise instructional sessions lead by a train exercise specialist. The exercise protocol focuses on improving balance, walking, lower limb and core muscle strength, and spasticity. The instructional session teaches participants a standardized series of exercises that focus on balance, muscle strength, and stretching. The exercises target lower limb & core muscle function. Once taught, participants will perform the exercises 3 times a week in their home as outlined in a manual. Subjects return in the first month and second month to ensure that exercises are being executed with correct form and appropriate intensity level. Compliance of at-home exercise will be assessed with diaries that participants complete every other week.
  Interventions: Behavioral: Home-based Exercise
- Control (No Intervention): Wait-list control.

INTERVENTIONS:
Behavioral: Home-based Exercise — This is a control group with no intervention
  Arms: Home-based Exercise

SUMMARY:
Over half of persons with multiple sclerosis (MS) report falling over a 6-month period and a majority of those who fall require medical attention for injuries. Importantly, balance dysfunction, muscle weakness, and spasticity are modifiable risk factors for falls among community-dwelling older adults and likely persons with MS. Indeed, there is evidence that these physiological risk factors can be minimized with exercise training in persons with MS and this might translate into a decrease in fall risk as documented in community-dwelling older adults.

The investigation will examine the effectiveness of a home-based exercise program that is designed to reduce fall risk by targeting specific fall risk factors including balance dysfunction and two of its latent causes, muscle weakness and spasticity in persons with multiple sclerosis. It is predicted that persons who receive home-based exercise program will have a reduction in fall risk.

DETAILED DESCRIPTION:
Over half of persons with multiple sclerosis (MS) report falling over a 6-month period and half of those who fall require medical attention for injuries. To make matters worse, a fall can result in activity curtailment, physiological deconditioning, and institutionalization. Importantly, balance dysfunction, muscle weakness, and spasticity are modifiable risk factors for falls among community-dwelling older adults and likely persons with MS. Indeed, there is evidence that these physiological risk factors can be minimized with exercise training in persons with MS and this might translate into a decrease in fall risk as documented in community-dwelling older adults. To that end, an appropriately designed exercise training program that targets specific, modifiable risk factors might be effective for decreasing the fall risk in persons with MS.

The investigation will examine the effectiveness of a home-based exercise program that is designed to reduce fall risk by targeting specific fall risk factors including balance dysfunction and two of its latent causes, muscle weakness and spasticity in persons with multiple sclerosis. It is predicted that persons who receive home-based exercise program will have a reduction in fall risk.

Participants will undergo multidimensional assessment of walking, balance, muscle strength, spasticity and fall risk prior to and immediately following the 12 week intervention. Following baseline assessment participants will be randomized into intervention or control groups. The intervention group will receive exercise instruction 4 times over 2 months. The home-based exercise protocol will focus on improving balance, walking, lower limb and core muscle strength, and spasticity, all potential determinants of falling.

ELIGIBILITY:
Inclusion Criteria:

* having an established definite diagnosis of MS;
* being independently ambulatory or ambulatory with an aid;
* having the visual ability necessary to read 14 point font;
* meeting the age requirement (i.e., 50-75 years of age);
* having fallen at least once in the past year and
* willingness and ability to attend the training sessions and testing sessions

Exclusion Criteria:

* non-ambulatory;
* risk factors contra-indicative for undertaking strenuous exercise as determined by the physical activity readiness questionnaire.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Physiological Fall risk | 3 months
  Physiological fall risk will be determined by the physiological profile assessment which assesses physiological function related to fall risk by combining measures of vision, proprioception, lower-limb strength, postural sway, and cognitive function.

SECONDARY OUTCOMES:
Mobility | 3 months
  Mobility will be quantified with performance on timed 25 foot walk (T25W), timed up and go (TUG), Six spot step test, 6 minute walk and the MS walking scale-12.
Balance | 3 Months
  Balance will be quantified with the Berg Balance scale; self-report of balance impairment (ABC); and force platform metrics (sway range and velocity).
Spasticity | 3 Months
  Spasticity will be assessed with the modified ashworth scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sosnoff, PhD, Principal Investigator — University of Illinois at UC
Locations (1):
- University of Illinois UC, Urbana, Illinois, United States

REFERENCES:
- [Result] Sosnoff JJ, Finlayson M, McAuley E, Morrison S, Motl RW. Home-based exercise program and fall-risk reduction in older adults with multiple sclerosis: phase 1 randomized controlled trial. Clin Rehabil. 2014 Mar;28(3):254-63. doi: 10.1177/0269215513501092. Epub 2013 Aug 27. PMID 23983091